CLINICAL TRIAL: NCT03807050
Title: Safety and Pharmacokinetics of Astaxanthin-Rich Carotenoid Extract (AstaFerm™) Administered as a Single Oral Dose to Healthy Adults
Brief Title: Safety and Pharmacokinetics of Phaffia Rhodozyma Astaxanthin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NextFerm Technologies LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AstaFerm 001
Record Dates: First submitted 2019-01-09; First posted 2019-01-16 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-01

CONDITIONS: Absorption; Chemicals
Keywords: Pharmacokinetics
MeSH Terms: interventions — astaxanthine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Astaxanthin (Experimental): Astaxanthin capsules containing 50 milligram astaxanthin derived from the yeast Phaffia rhodozyma (Xanthophyllomyces dendrorhous)
  Interventions: Dietary Supplement: Astaxanthin

INTERVENTIONS:
Dietary Supplement: Astaxanthin — Capsules containing astaxanthin derived from the yeast Phaffia rhodozyma .
  Other Names: AstaFerm

SUMMARY:
Astaxanthin is a xanthophyll carotenoid, a naturally occurring lipid-soluble red pigment. Apart from its coloring ability it is also a strong antioxidative ingredient and contains health-promoting properties.

Study aim is to monitor the safety and tolerability of AstaFerm™, an astaxanthin dietary supplement derived from the yeast Phaffia rhodozyma. Pharmacokinetics profile is tested in 12 healthy male adults who received a single dose of AstaFerm™ in a single-center, open-label, non-randomized, single-dose study. Subjects are admitted to the clinical research center on the evening before dosing. On the next morning, after overnight fast, pre-dosing plasma sampling is performed, then they receive a fat balanced breakfast followed by a single administration of AstaFerm™ capsules. The capsules contain 50 milligram astaxanthin derived from Phaffia rhodozyma. Following dosing, blood sampling is performed for 24 hours in-house (2, 4, 6, 8, 10, 12 and 24-hours post-dose) and ambulatory at 48, 72- and 168-hours post-dose. Blood for antioxidant activity assessment is also drawn.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male volunteers between 18 and <46 years of age.
2. Subjects who provide written informed consent to participate in the study.
3. BMI ranging from 18.0 to <30.0, calculated as Weight (Kg)/Height (m2).
4. Non-smoking (by declaration) for a period of at least 6 months.
5. No known history of significant neurological, renal, cardiovascular (including known structural cardiac abnormalities or hypertension), respiratory (asthma), endocrine, gastrointestinal, hepatic or hematopoietic disease, neoplasm, psychiatric or any other clinically significant medical disorder, which in the investigator's judgment contraindicate administration of the study medications.
6. No history of drug or alcohol abuse.
7. No known allergy or hypersensitivity to any drug or food.
8. No clinically significant abnormalities in screening physical exam.
9. No clinically significant abnormalities in clinical laboratory parameters (hematology, biochemistry and urinalysis) at Screening, as determined by the study physicians.
10. Negative HIV antibody, Hepatitis B surface antigen and Hepatitis C antibody tests at Screening.
11. No significant abnormalities in electrocardiogram.at Screening.
12. Subjects with negative urinary drugs of abuse screen determined at Screening and on admission to the clinical research center prior to dosing day.
13. Subjects must be able to adhere to the visit schedule and protocol requirements and be available to complete the study.
14. Subjects must satisfy a medical examiner about their fitness to participate in the study.

Exclusion Criteria:

1. Subjects with any clinically significant abnormality upon physical examination or in the clinical laboratory test values.
2. Subjects with a history of clinically defined peptic ulcer or any gastrointestinal surgery other than appendectomy or herniotomy, or with any gastrointestinal disorder likely to influence supplement absorption, or with any history of severe gastrointestinal narrowing, or frequent nausea or emesis, regardless of etiology.
3. Subjects with significant allergic response to any drug or history of food allergies deemed clinically significant or exclusionary for the study.
4. Adherence (for whatever reason) to an abnormal diet during the 4 weeks prior to the study, or subjects with recent significant change in body weight.
5. Treatment with prescription or over-the-counter drugs, nutraceuticals including vitamins, herbal medications, food supplements and other prescription drugs not mentioned above, within 7 days prior to first dosing day.
6. Use of paracetamol (acetaminophen) less than 24 hours before the first dosing day.
7. Subjects who donated blood or received blood or plasma derivatives in the three months preceding the first study dosing.
8. Participation in another clinical trial with drugs within 3 months prior to first study dosing day (calculated from the previous study's last dosing date).
9. Subjects with an inability to communicate well with the investigators and Clinical research Center staff (i.e., language problem, poor mental development or impaired cerebral function).
10. Subjects that have difficulty fasting or consuming the standard meals that will be provided.
11. Subjects with any acute medical situation (e.g. acute infection) within 48 hours of study start, which is considered of significance by the Principal Investigator.
12. Subjects who are non-cooperative or unwilling to sign the consent form.

Ages: 18 Years to 46 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2018-12-23 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Cmax | Estimated to be at 8 to 10 hours after dosing
  The maximum plasma concentration obtained in average of 12 subjects
AUC 0-t | 168 hours after dosing
  Calculate Area under the plasma concentration versus time curve from time =0 h to time of the last measurable concentration of 12 subjects
Time max | Estimated to be at 8 to 10 hours after dosing
  Time at which Cmax occurs

SECONDARY OUTCOMES:
Adverse Events (AEs) | 15 days
  Number of subjects that reported incidence of adverse events and details of adverse events that were reported

CONTACTS AND LOCATIONS:
Overall Officials: Oren Shibolet, Prof., Principal Investigator — Tel Aviv Sourasky Medical Center Israel
Locations (1):
- Sourasky Medical Center, Tel Aviv, Israel